CLINICAL TRIAL: NCT01182818
Title: FASEP Fabry and Stroke Epidemiological Protocol RISK FACTORS IN ISCHEMIC STROKE PATIENTS WITH FABRY DISEASE AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Fabry and Stroke Epidemiological Protocol (FASEP): Risk Factors In Ischemic Stroke Patients With Fabry Disease
Acronym: FASEP
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Prof. Dr. Arndt Rolfs, Prof. Dr. med., University of Rostock
Other Study IDs: FD01/2010
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cerebrovascular Accident; Stroke, Acute; Cerebral Stroke
Keywords: Cerebrovascular Accident; Cerebrovascular Accident, Acute; Fabry Disease; Fabry´s Disease; Anderson-Fabry Disease; CVA (Cerebrovascular Accident); Stroke, Acute; Cerebral Stroke
MeSH Terms: conditions — Stroke; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fabry diagnostic will be done centrally: blood samples will be stored for analysis of a-galactosidase in blood, Gb3 as well as lyso-Gb3. In all cases direct analysis of the gene will be done, especially in females where due to the Lyonisation effect a-galactosidase activity might be normal in blood although the patient might suffer from Fabry disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: all adult patients (18 - 60 years of age) with an acute cerebrovascular event of any etiology

SUMMARY:
More than one million people in Europe suffer from a stroke every day. Normally older people have a stroke, but also a significant number of younger people between 18 and 55 years. Usually, these can only be explained for a minority by the classical risk factors such as diabetes, overweight and high blood pressure. New studies indicate that in about 1 - 2 % of the younger stroke patients the etiology can be an undiagnosed genetic disease, e.g. Fabry disease. Fabry disease is a lysosomal storage disorder known to cause vasculopathy. The purpose of this study is to determine in a large number of young stroke patients, how many strokes were caused by Fabry disease and what risk factors might be able to predict this disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 - 60 years of age) with an acute ischemic cerebrovascular event either acute ischemic stroke or transient ischemic attack within 10 days
* Diagnosis of the cerebrovascular event (CVE) by a stroke experienced physician
* Diagnostic procedures for CVE according to the local guidelines and recommendations
* Written informed consent from patient or legal representative according to local regulations

Exclusion Criteria:

* Patients being younger than 18 years or older than 60 years of age.
* Acute ischemic stroke or transient ischemic attack longer than 10 days before enrollment into the study
* CVE associated with intracranial hemorrhage as evidenced by cerebral CT scan
* Any uncertainty in the diagnosis
* No written informed consent from the patient or legal representative

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with acute ischemic cerebrovascular event of any ischemic etiology
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, MD, Principal Investigator — University of Rostock, Albrecht-Kossel-Institute for Neuroregeneration
Locations (14):
- Germany (13):
  - Department of Neurology, Kreiskrankenhaus Altenburg, Altenburg
  - Dept. of Neurology, Vivantes Netzwerk für Gesundheit GmbH, Klinikum Neukölln, Berlin
  - Department of Neurology, Allgemeines Krankenhaus Celle, Celle
  - Department of Neurology, Klinikum Chemnitz gGmbH, Chemnitz
  - Heinrich-Heine University Duesseldorf, Dept. of Neurology, Düsseldorf
  - Universitätsklinikum Giessen, Department of Neurology, Giessen
  - Department of Neurology S10, Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universität Heidelberg, Klinik für Neurologie, Heidelberg
  - Department of Neurology, Universitaetsklinikum Jena, Jena
  - Dept. of Neurology, Ökumenisches Hainich Klinikum gGmbH, Mühlhausen / Thürigen
  - Universitätsklinikum Regensburg, Klinik für Neurologie, Regensburg
  - University of Rostock, Department of Neurology, Rostock
  - University of Ulm, Department of Neurology, Ulm
- Institute of Psychiatry and Neurology, Dept. of Neurology, Warsaw, Poland

REFERENCES:
- See also: study homepage — http://www.fasep.eu